CLINICAL TRIAL: NCT02245386
Title: Effects of Pregnancy and Parturition on Pelvic Floor Morphology and Sexual Function in Egyptian Women.
Brief Title: Effects of Pregnancy and Childbirth on Pelvic Floor Morphology and Sexual Function in Egyptian Women
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Muhamed Osman, Dr, Al-Azhar University
Other Study IDs: 1781956
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Pregnancy, Childbirth and Puerperal Disorders
MeSH Terms: conditions — Puerperal Disorders

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group 1: (40 women after normal vaginal delivery) submitted to transperineal pelvic floor ultrasound 48-72 hours postpartum.
  Interventions: Radiation: transperineal pelvic floor ultrasound
- Group 2: (40 women after urgent cesarean section) submitted to transperineal pelvic floor ultrasound 48-72 hours postpartum.
  Interventions: Radiation: transperineal pelvic floor ultrasound
- Group 3: (40 women after elective cesarean section) submitted to transperineal pelvic floor ultrasound 48-72 hours postpartum.
  Interventions: Radiation: transperineal pelvic floor ultrasound

INTERVENTIONS:
Radiation: transperineal pelvic floor ultrasound — Transperineal pelvic floor ultrasound applied for the submitted 120 women "primiparae" (40 women after normal vaginal delivery), (40 women after urgent cesarean section), (40 women after elective cesarean section), in early postpartum period (48 to 72) hours postpartum, to evaluate levator ani morphology.

SUMMARY:
To evaluate levator ani muscle morphology following normal vaginal delivery and cesarean section (elective and emergent), using three-dimensional (3D) transperineal ultrasound, and to study the effect of mode of delivery on female sexual function.

DETAILED DESCRIPTION:
1. transperineal pelvic floor ultrasound applied for the submitted 120 women "primiparae" (40 women after normal vaginal delivery), (40 women after urgent cesarean section), (40 women after elective cesarean section), in early postpartum period (48 to 72) hours postpartum, to evaluate levator ani morphology.
2. answering of the validated female sexual function index (F.S.F.I) three months postpartum period for same cases submitted to ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* primiparae in early postpartum period (48 hours to72 hours). written consent was taken. easy communicable, reachable women for further requirements.

Exclusion Criteria:

1. Refused consent.
2. Previous vaginal or cesarean delivery.
3. Severe mental illness.
4. Severe physical handicap or difficulties in communication.
5. Women without postpartum active sexual life or separate from their spouse.
6. Past history of sexual dysfunction.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primiparae in early postpartum period (48 hours to72 hours). written consent was taken. easy communicable, reachable women for further requirements.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle strength as assessed by three/four dimensional translabial pelvic floor ultrasound | early postpartum period (48 to 72) hours postpartum
Sexual function of pelvic floor as assessed by the validated female sexual function index | at 3 months after delivery

SECONDARY OUTCOMES:
Trauma or avulsion of levator ani muscle as assessed by three/four dimensional translabial pelvic floor ultrasound | 6 months after delivery.
Sexual function as assessed by the validated female sexual function index | 3 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Muhamed Osman, Ms, Principal Investigator — Al-Azhar University